CLINICAL TRIAL: NCT04536935
Title: Acceptability, Usability and Effectiveness of Mental Health Apps for Suicide Prevention in Essential Workers and the Unemployed During SARS-CoV-2
Brief Title: Mobile Mental Health Apps for Suicide Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kate Comtois, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010842; 5P50MH115837-03 (NIH)
Record Dates: First submitted 2020-08-22; First posted 2020-09-03 (Actual); Results first posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Depression; Anxiety; Emotional Regulation
MeSH Terms: conditions — Depression; Anxiety Disorders; Emotional Regulation | interventions — Calmodulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 2: Mobile Mental Health App - 1 (Active Comparator): Participants randomized to a free mobile mental health application that focuses on meditation.
  Interventions: Behavioral: Mobile Mental Health App - 1
- Phase 2: Mobile Mental Health App - 2 (Active Comparator): Participants randomized to a free mobile mental health application that assists with coping with COVID-19.
  Interventions: Behavioral: Mobile Mental Health App - 2
- Phase 2: Mobile Mental Health App - 3 (Active Comparator): Participants randomized to a free mobile mental health application that focuses on positive psychology.
  Interventions: Behavioral: Mobile Mental Health App - 3
- Phase 2: Mobile Mental Health App - 4 (Active Comparator): Participants randomized to a free mobile application that addresses mental health issues through mood tracking.
  Interventions: Behavioral: Mobile Mental Health App - 4

INTERVENTIONS:
Behavioral: Mobile Mental Health App - 1 — Free mobile mental health application that focuses on meditation
  Other Names: Calm
  Arms: Phase 2: Mobile Mental Health App - 1
Behavioral: Mobile Mental Health App - 2 — Free mobile mental health application that assists with coping with COVID-19
  Other Names: COVID Coach
  Arms: Phase 2: Mobile Mental Health App - 2
Behavioral: Mobile Mental Health App - 3 — Free mobile mental health application that focuses on positive psychology.
  Other Names: 7 Cups of Tea
  Arms: Phase 2: Mobile Mental Health App - 3
Behavioral: Mobile Mental Health App - 4 — Free mobile application that addresses mental health issues through mood tracking
  Other Names: Beautiful Mood
  Arms: Phase 2: Mobile Mental Health App - 4

SUMMARY:
Access to mental health care by essential workers and the unemployed during the COVID19 pandemic has been challenging. Usual access to mental health care is limited by social distancing, and for many now unemployed due to closures of businesses, insurance is insufficient to cover the costs of mental health care. For these individuals who are at risk for suicide (isolation, unemployment, financial crisis plus past suicide attempts, significant mental health challenges), access to care is crucial and many maybe turning to online and accessible interventions, such as mental health apps and other online resources. Indeed, organizations such as the VA have already created free access mobile applications for mental health in anticipation of this need. Using Psyberguide, the investigators will identify the top ten free apps that address mental health issues and conduct a nation-wide evaluation of these apps with participants who are essential workers and unemployed with risk for suicide. Participants will first be surveyed about which strategies they have used to manage mental health issues, what apps and online tools they have used, and what usability challenges they have faced. The investigators will then ask a random sample of participant to engage in a randomized trial of these top-rated apps for 4 weeks. Apps will be rated on usability, acceptability, feasibility and effectiveness. Results from this trial will be quickly disseminated through several avenues: (1) the UWAC website and ALACRITY Centers network; (2) through CREATIV Lab's partnership with Mental Health America; (3) through the UW Center for Suicide Prevention and Recovery (CSPAR) and partnerships with other suicide focused organizations including Forefront, the American Foundation for Suicide Prevention, that American Association of Suicidology, the Rocky Mountain MIRECC, and the Defense Suicide Prevention Office and (4) through local partnership with King County and WA state contact tracers.

DETAILED DESCRIPTION:
Participants will be recruited nationally via Prolific. Investigators will aim to recruit 1,000 participants in the clinical trial who are essential workers and/or unemployed due to COVID-19 and have a past history of mental health issues or experiencing suicide ideation motivational risk factors to be randomized (250 per group) to one of the four apps. They will be asked to download their assigned app and use it for 4 weeks. After 4 weeks of use, participants will be asked to provide an evaluation of acceptability, feasibility and usability of the app, how often they used the app, and if they found the app helpful. Participants will also be asked to complete clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* 19 years old and older
* Identify as an essential worker or unemployed due to COVID-19
* English-speaking
* Access to a mobile device (e.g. smartphone or tablet)
* Based in the United States

Phase 2

* 19 years old and older
* Scored at or above validated cut off scores in Phase 1 (PHQ-2>3; GAD-2>3; SBQ-R>7) or reported history of past suicide attempt
* Identify as an essential worker or unemployed due to COVID-19
* English-speaking
* Access to a mobile device (e.g. smartphone or tablet)
* Based in the United States

Exclusion Criteria:

Phase 1

* Under the age of 19
* Neither an essential worker nor unemployed due to COVID-19
* Non-English speaking
* No access to a mobile device (e.g. smartphone or tablet)
* Not based in the United States

Phase 2

* Under the age of 19
* Did not score at or above validated cut off scores in Phase 1 (PHQ-2>3; GAD-2>3; SBQ-R>7) nor reported history of past suicide attempt
* Neither an essential worker nor unemployed due to COVID-19
* Non-English speaking
* No access to a mobile device (e.g. smartphone or tablet)
* Not based in the United States

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 838 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Comtois KA, Mata-Greve F, Johnson M, Pullmann MD, Mosser B, Arean P. Effectiveness of Mental Health Apps for Distress During COVID-19 in US Unemployed and Essential Workers: Remote Pragmatic Randomized Clinical Trial. JMIR Mhealth Uhealth. 2022 Nov 7;10(11):e41689. doi: 10.2196/41689. PMID 36191176
- [Derived] Mata-Greve F, Johnson M, Blanchard BE. A longitudinal examination of cultural risk factors of suicide and emotion regulation. Am J Orthopsychiatry. 2022;92(5):635-645. doi: 10.1037/ort0000629. Epub 2022 May 26. PMID 35617246

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Investigators will aim to recruit 1,000 participants in the clinical trial who are essential workers and/or unemployed due to COVID-19 and have a past history of mental health issues or experiencing suicide ideation motivational risk factors to be randomized (250 per group) to one of the four apps.
Groups:
- Phase 2: Mobile Mental Health App - 1 - Calm: Mobile Mental Health App - 1: Free mobile mental health application that focuses on meditation
- Phase 2: Mobile Mental Health App - 2 - COVID Coach: Mobile Mental Health App - 2: Free mobile mental health application that assists with coping with COVID-19
- Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea: Mobile Mental Health App - 3: Free mobile mental health application that focuses on positive psychology.
- Phase 2: Mobile Mental Health App - 4 - Beautiful Mood: Mobile Mental Health App - 4: Free mobile application that addresses mental health issues through mood tracking
Period: RCT Baseline
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Started | 204 | 212 | 209 | 213
Completed | 204 | 212 | 209 | 213
Not Completed | 0 | 0 | 0 | 0
Period: RCT Follow-Up
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Started | 204 | 212 | 209 | 213
Completed | 155 | 168 | 152 | 168
Not Completed | 49 | 44 | 57 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood | Total
Number analyzed (Participants) | 204 | 212 | 209 | 213 | 838
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant did not provide age information.
  years
    number analyzed (Participants) | 204 | 212 | 208 | 213 | 837
    (all) | 31.4 (10.0) | 29.9 (8.2) | 31.4 (9.4) | 31.8 (10.1) | 31.1 (9.5)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: A total of five participants did not provide gender data.
  Participants
    Gender: number analyzed (Participants) | 204 | 209 | 208 | 212 | 833
    Gender: Women | 118 | 118 | 115 | 116 | 467
    Gender: Gender Diverse | 1 | 1 | 2 | 0 | 4
    Gender: Men | 78 | 80 | 83 | 85 | 326
    Gender: Non-binary | 7 | 7 | 7 | 10 | 31
    Gender: Transgender | 0 | 3 | 1 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 17 | 19 | 23 | 80
  Not Hispanic or Latino | 183 | 190 | 189 | 188 | 750
  Unknown or Not Reported | 0 | 5 | 1 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 0 | 3 | 8
  Asian | 26 | 23 | 13 | 22 | 84
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 20 | 12 | 15 | 58
  White | 149 | 142 | 169 | 156 | 616
  More than one race | 10 | 18 | 12 | 13 | 53
  Unknown or Not Reported | 5 | 7 | 3 | 4 | 19
Marital Status [Count of Participants; unit: Participants] — Population: Nine participants did not provide marital status data.
  Participants
    number analyzed (Participants) | 203 | 209 | 207 | 210 | 829
    Divorced | 10 | 11 | 17 | 14 | 52
    Married (including same sex partnership) | 56 | 56 | 61 | 61 | 234
    Never marred | 131 | 136 | 123 | 134 | 524
    Separated | 4 | 6 | 3 | 1 | 14
    Widowed | 2 | 0 | 3 | 0 | 5
Education [Count of Participants; unit: Participants] — Population: One participant did not provide education data.
  Participants
    number analyzed (Participants) | 204 | 211 | 209 | 213 | 837
    High School GED, or less | 27 | 28 | 23 | 22 | 100
    Some college | 54 | 50 | 51 | 74 | 229
    Trade/Technical/Vocational | 25 | 27 | 32 | 19 | 103
    Bachelor's Degree | 65 | 73 | 67 | 64 | 269
    Higher Education | 33 | 33 | 36 | 34 | 136
Income [Count of Participants; unit: Participants] — Population: A total of ten participants did not provide income data.
  Participants
    number analyzed (Participants) | 203 | 206 | 207 | 212 | 828
    Below $10K | 31 | 37 | 30 | 30 | 128
    $10,000 - $31,199 | 58 | 56 | 53 | 60 | 227
    $31,200 - $33,280 | 5 | 17 | 8 | 17 | 47
    $33,281 - $49,999 | 31 | 31 | 31 | 29 | 122
    $50,000 - $59,999 | 23 | 16 | 17 | 11 | 67
    $60,000 - $69,999 | 14 | 10 | 14 | 10 | 48
    $70,000 - $99,999 | 20 | 19 | 27 | 34 | 100
    $100,000 - $149,999 | 11 | 15 | 14 | 14 | 54
    $150,000 or above | 10 | 5 | 13 | 7 | 35

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) consists of 9 depression items and one disability item. Each item is associated with a DSM symptom of depression, which the participant rates whether or not they have experienced the symptom over the last two weeks, with severity rating of 0-3. It is one of the few measures that is brief (it takes less than one minute to give) and has been found to have excellent sensitivity to change over time, with a total sum score ranging from 0 - 27. Higher scores indicate higher depression symptom severity.
Time Frame: PHQ-9 at RCT baseline and RCT follow-up; duration of 4 weeks.
Population: Participants providing both RCT baseline and RCT follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - Covid Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 155 | 166 | 151 | 165
score on a scale
  RCT Baseline | 10.1 (5.7) | 11.2 (6.3) | 11.0 (6.5) | 10.6 (6.6)
  RCT Follow-Up | 8.5 (5.9) | 9.8 (6.7) | 9.7 (6.6) | 9.1 (6.5)
Statistical Analysis 1: Comparison: Phase 2: Mobile Mental Health App - 1 - Calm vs Phase 2: Mobile Mental Health App - 2 - Covid Coach vs Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea vs Phase 2: Mobile Mental Health App - 4 - Beautiful Mood; Test type: Superiority — A series of mixed effects models using restricted maximum likelihood estimation were built to test linear time change on the PHQ-9 and to test for condition differences at follow-up and change slope. Models were built in an outwardly nested fashion, such that an initial null model was computed, followed by models that added a random intercept, random time component, condition assignment, and condition x time interaction effects; p < .001, Mixed Models Analysis; Slope = -1.5, 95% CI 2-sided [-1.8 to -1.1], Standard Error of Mean 0.2

2. Primary Outcome: Generalized Anxiety Disorder (7-Item) Scale (GAD-7)
Description: The Generalized Anxiety Disorder Scale (GAD-7) is a 7- item screener for generalized anxiety. It consists of items related to generalized anxiety disorder. Participants rate on a scale of 0-3 how much they have experienced in the last two weeks to crease a total sum score ranging from 0 - 21. The scale is a valid screener for generalized anxiety symptoms. Higher scores indicate higher anxiety symptom severity.
Time Frame: GAD-7 at RCT baseline and RCT follow-up; duration of 4 weeks.
Population: Participants providing both RCT baseline and RCT follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 153 | 168 | 151 | 167
score on a scale
  RCT Baseline | 7.9 (4.8) | 9.2 (5.6) | 8.9 (5.6) | 8.8 (5.7)
  RCT Follow-Up | 6.7 (5.1) | 7.8 (5.6) | 7.3 (5.8) | 7.8 (5.6)
Statistical Analysis 1: Comparison: Phase 2: Mobile Mental Health App - 1 - Calm vs Phase 2: Mobile Mental Health App - 2 - COVID Coach vs Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea vs Phase 2: Mobile Mental Health App - 4 - Beautiful Mood; Test type: Other — A series of mixed effects models using restricted maximum likelihood estimation were built to test linear time change on the GAD-7 and to test for condition differences at follow-up and change slope. Models were built in an outwardly nested fashion, such that an initial null model was computed, followed by models that added a random intercept, random time component, condition assignment, and condition x time interaction effects; p < .001, Mixed Models Analysis; Slope = -1.3, 95% CI 2-sided [-1.6 to -1.0], Standard Error of Mean 0.2

3. Primary Outcome: Brief Difficulties With Emotional Regulation Scale (DERS)
Description: The Brief Difficulties with Emotional Regulation Scale (DERS) is a brief, 36-item, self-report questionnaire designed to assess multiple aspects of emotion dysregulation. a 36-item self-report measure of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Total scores range from 18 - 90 with higher scores indicate more difficulty in emotion regulation.
Time Frame: DERS at RCT baseline and RCT follow-up; duration of four weeks.
Population: Participants providing both RCT baseline and RCT follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 153 | 163 | 148 | 165
score on a scale
  RCT Baseline | 42.8 (11.7) | 44.6 (12.5) | 44.6 (12.8) | 44.5 (13.0)
  RCT Follow-Up | 42.2 (13.1) | 44.6 (14.0) | 44.9 (13.0) | 44.6 (14.2)
Statistical Analysis 1: Comparison: Phase 2: Mobile Mental Health App - 1 - Calm vs Phase 2: Mobile Mental Health App - 2 - COVID Coach vs Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea vs Phase 2: Mobile Mental Health App - 4 - Beautiful Mood; Test type: Other — A series of mixed effects models using restricted maximum likelihood estimation were built to test linear time change on the DERS and to test for condition differences at follow-up and change slope. Models were built in an outwardly nested fashion, such that an initial null model was computed, followed by models that added a random intercept, random time component, condition assignment, and condition x time interaction effects; p = .73, Mixed Models Analysis

4. Primary Outcome: Suicidal Behavioral Questionnaire-Revised (SBQ-R)
Description: The suicidal behavioral questionnaire revised (SBQ-R) is a self-report questionnaire designed to identify risk factors for suicide. Total scores range from 3 to 18, with higher scores indicate indicating higher risk of suicidal behavior.
Time Frame: SBQ-R RCT baseline and RCT follow-up; duration of four weeks.
Population: Participants providing both RCT baseline and RCT follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 144 | 159 | 139 | 154
score on a scale
  RCT Baseline | 6.6 (3.3) | 6.9 (3.8) | 7.1 (3.9) | 7.1 (3.6)
  RCT Follow-Up | 6.4 (3.3) | 6.7 (3.7) | 7.1 (3.9) | 7.0 (3.8)
Statistical Analysis 1: Comparison: Phase 2: Mobile Mental Health App - 1 - Calm vs Phase 2: Mobile Mental Health App - 2 - COVID Coach vs Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea vs Phase 2: Mobile Mental Health App - 4 - Beautiful Mood; Test type: Other; p = .25, Mixed Models Analysis

5. Secondary Outcome: Acceptability of Intervention Measure (AIM)
Description: This is a four item measure of intervention acceptability, where each item is rated on a 1-5 scale, with 1 = not at all acceptable and 5 = very acceptable. Total mean scores range from 1 - 5, with higher scores indicating higher acceptability. Participants will complete this measure after 4 weeks of using the mobile mental health app to which they are randomized.
Time Frame: Participants will complete this measure at RCT Follow-Up; after 4 weeks of using the mobile mental health app to which they are randomized.
Population: Participants providing AIM usability data at RCT Follow-Up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 152 | 164 | 150 | 165
score on a scale | 3.4 (1.0) | 3.6 (0.9) | 3.4 (1.0) | 3.5 (1.0)
Statistical Analysis 1: Comparison: Phase 2: Mobile Mental Health App - 1 - Calm vs Phase 2: Mobile Mental Health App - 2 - COVID Coach vs Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea vs Phase 2: Mobile Mental Health App - 4 - Beautiful Mood; Test type: Superiority; p = .22, ANOVA

6. Secondary Outcome: Intervention Appropriateness Measure (IAM)
Description: This is a four item measure of intervention appropriateness, where each item is rated on a 1-5 scale, with 1 = not at all acceptable and 5 = very acceptable. A total mean score ranges from 1 - 5, with higher scores indicating higher appropriateness. Participants will complete this measure after 4 weeks of using the mobile mental health app to which they are randomized.
Time Frame: as for outcome 5
Population: Participants providing IAM usability data at RCT Follow-Up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 152 | 166 | 152 | 162
score on a scale | 3.6 (0.9) | 3.7 (0.9) | 3.6 (0.9) | 3.7 (0.8)
Statistical Analysis 1: Comparison: Phase 2: Mobile Mental Health App - 1 - Calm vs Phase 2: Mobile Mental Health App - 2 - COVID Coach vs Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea vs Phase 2: Mobile Mental Health App - 4 - Beautiful Mood; Test type: Superiority; p = .48, ANOVA

7. Secondary Outcome: Intervention Usability Scale (IUS)
Description: The Intervention Usability Scale (IUS) is a 10-item measure that assesses intervention usability through its likeability, learnability, difficulty, need for support, system integration, and efficiency. The measure is based on the System Usability Scale (SUS), a standardized, normed measure in industry for digital tools. Total scores can range from 0 - 100 with higher scores indicate higher levels of usability.
Time Frame: as for outcome 5
Population: Participants contributing IUS data at RCT Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 155 | 167 | 152 | 166
score on a scale | 66.8 (17.3) | 71.2 (15.4) | 65.2 (17.7) | 72.9 (16.7)
Statistical Analysis 1: Comparison: Phase 2: Mobile Mental Health App - 1 - Calm vs Phase 2: Mobile Mental Health App - 2 - COVID Coach vs Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea vs Phase 2: Mobile Mental Health App - 4 - Beautiful Mood; Test type: Superiority; p < .0001, ANOVA

8. Secondary Outcome: Feasibility of Intervention Measure (FIM)
Description: This is a four item measure of intervention feasibility, where each item is rated on a 1-5 scale, with 1 = not at all acceptable and 5 = very acceptable, with a total mean score ranging from 1 to 5. Participants will complete this measure after 4 weeks of using the mobile mental health app to which they are randomized. High scores indicate higher levels of feasibility. No data displayed because outcome measure data was not collected therefore zero total participants analyzed.
Time Frame: as for outcome 5
Population: No data displayed because outcome measure has zero total participants analyzed.
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Other Pre Specified Outcome: PARS EQ-5D
Description: Standardized measure of health status with a total score range of 0 - 1. Maximum score of one indicates the best health state.
Time Frame: PARS EQ-5D at RCT baseline and RCT follow-up; duration of 4 weeks.
Population: Participants providing both RCT baseline and RCT follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 153 | 167 | 150 | 165
score on a scale
  RCT Baseline | 0.8 (0.1) | 0.7 (0.2) | 0.8 (0.2) | 0.8 (0.1)
  RCT Follow-Up | 0.8 (0.1) | 0.8 (0.2) | 0.8 (0.2) | 0.8 (0.1)

10. Other Pre Specified Outcome: CAGE-AID
Description: Standardized measure of alcohol/drug use with a total score range of 0 - 4. Higher scores indicate higher risk for substance use.
Time Frame: Participants will complete the CAGE-AID at RCT follow-up; after 4 weeks of using the mobile mental health app to which they are randomized.
Population: Participants contributing to CAGE-AID data at RCT follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 152 | 162 | 146 | 160
score on a scale | 0.9 (1.4) | 1.0 (1.4) | 1.3 (1.5) | 1.2 (1.5)

11. Other Pre Specified Outcome: Brief Resilience Scale (BRS)
Description: The Brief Resilience Scale (BRS) is a 6-item, self-reported measure of an individual's ability to bounce back, resist illness, adapt to stress, or thrive in the face of adversity. Responses for all 6 items are on a scale of 1-5, with a total mean score ranging from 1 to 5. Higher score indicates higher resilience.
Time Frame: Participants will complete the BRS at RCT follow-up; after 4 weeks of using the mobile mental health app to which they are randomized.
Population: Participants contributing BRS data at RCT follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 155 | 168 | 151 | 166
score on a scale | 2.9 (0.9) | 3.0 (0.9) | 3.0 (0.9) | 3.0 (1.0)

12. Other Pre Specified Outcome: Defeat Scale
Description: Gilbert and Allan (1998) designed the items on this scale in order to depict a sense of failed struggle and losing rank. This measure requests participants to respond to 16 items on a 5-point Likert scale (ranging from 0 = 'Never' to 4 = 'Always') asking them how much they had felt defeated in the previous seven days, for example item 1 'I feel that I have not made it in life'. This scale has very high internal consistency with Alpha coefficients of 0.94 for females and 0.93 for males in both groups, furthermore reliability of 0.94 for students and 0.93 for depressed group. Total score can range from 0 to 64. Higher scores indicate higher levels of defeat.
Time Frame: Participants will complete the Defeat Scale at RCT follow-up; after 4 weeks of using the mobile mental health app to which they are randomized.
Population: Participants contributing Defeat Scale data at RCT follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 155 | 167 | 152 | 167
score on a scale | 28.6 (15.4) | 29.5 (15.2) | 28.8 (15.2) | 27.4 (16.3)

13. Other Pre Specified Outcome: Entrapment Scale
Description: This 16-item entrapment scale asks participants to indicate on a 5-point scale the degree to which the items represent their thoughts and feelings. The response options are 0 = 'not at all like me', 1 = 'a little bit like me', 2 = 'moderately like me', 3= 'quite a bit like me' and 4 = 'extremely like me'. Gilbert and Allan (1998) reported high levels of internal consistency for both student and depressed groups, with Cronbach's alphas respectively of .93 and .86 in Internal Entrapment, and .88 and .89 in External Entrapment. Total score can range from 0 to 64. Higher scores indicate higher levels of entrapment.
Time Frame: Participants will complete the Entrapment Scale at RCT follow-up; after 4 weeks of using the mobile mental health app to which they are randomized.
Population: Participants contributing entrapment data at RCT follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 154 | 168 | 152 | 167
score on a scale | 20.6 (15.1) | 23.2 (16.7) | 22.8 (16.7) | 21.7 (16.7)

14. Other Pre Specified Outcome: Interpersonal Needs Questionnaire
Description: Brief questionnaire that asks respondents to think about themselves and other people, based on the respondent's current beliefs and experiences. Higher scores indicate higher levels of thwarted belongingness (subscale range 9 to 63) and perceived burdensomeness (subscale range 9 to 63).
Time Frame: Participants will complete the Interpersonal Needs Questionnaire at RCT follow-up; after 4 weeks of using the mobile mental health app to which they are randomized.
Population: Participants contributing to interpersonal needs data at RCT follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 155 | 168 | 152 | 168
score on a scale
  Thwarted Belongingness: number analyzed (Participants) | 155 | 166 | 152 | 168
  Thwarted Belongingness | 30.8 (13.5) | 32.3 (12.4) | 32.8 (13.3) | 30.3 (13.1)
  Perceived Burdensomeness: number analyzed (Participants) | 154 | 168 | 152 | 167
  Perceived Burdensomeness | 22.8 (12.9) | 25.7 (13.8) | 25.1 (13.7) | 23.4 (13.6)

15. Other Pre Specified Outcome: Loneliness and Social Distress Scale
Description: No data displayed because outcome measure data was not collected therefore zero total participants analyzed.
Time Frame: Loneliness and Social Distress Scale at 4 weeks
Population: No data displayed because outcome measure has zero total participants analyzed.
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Phase 2: Mobile Mental Health App - 1 - Calm | Phase 2: Mobile Mental Health App - 2 - COVID Coach | Phase 2: Mobile Mental Health App - 3 - 7 Cups of Tea | Phase 2: Mobile Mental Health App - 4 - Beautiful Mood
All-Cause Mortality (participants affected / at risk) | 0/204 | 0/212 | 0/209 | 0/213
Serious Adverse Events (participants affected / at risk) | 0/204 | 0/212 | 0/209 | 0/213
Other Adverse Events (participants affected / at risk) | 0/204 | 0/212 | 0/209 | 0/213

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT04536935/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT04536935/ICF_001.pdf